CLINICAL TRIAL: NCT06386159
Title: Clinical Application of Comprehensive Intervention Scheme for Post-extubation Dysphagia Based on Neuroregulatory Mechanism
Brief Title: Clinical Application of Comprehensive Intervention for PED Based on Neuroregulatory Mechanism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Jinhua Municipal Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-1178
Record Dates: First submitted 2024-04-24; First posted 2024-04-26 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-03

CONDITIONS: Post-extubation Dysphagia
Keywords: post-extubation dysphagia, electrical stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): During routine medical care and nursing, the responsible nurse provides daily oral care and delivers health education to patients and their caregivers regarding diet and swallowing safety. Within 8 hours after the removal of the endotracheal tube, the Standardized Swallowing Assessment (SSA) is used to screen for swallowing function. Patients are guided in food selection based on the severity of their swallowing difficulties and personal preferences, and are supplemented with enteral or parenteral nutrition or prescribed specific diets as directed by their doctor.
- Comprehensive Intervention Group (Active Comparator): On the basis of the control group, a comprehensive intervention plan determined through Delphi expert consultation is implemented for PED patients. This plan includes multidisciplinary collaboration, screening and assessment, oral sensory training, oral motor training, respiratory training, and feeding management. The duration and frequency of the exercises are tailored to the patient's actual condition.
  Interventions: Other: Comprehensive Intervention or Comprehensive Intervention Combined with Electrical vagus nerve stimulation
- Comprehensive Intervention Combined with Vagus Nerve Stimulation Group (Experimental): On the basis of the control group, a comprehensive intervention is implemented in combination with vagus nerve electrical stimulation.
  Interventions: Other: Comprehensive Intervention or Comprehensive Intervention Combined with Electrical vagus nerve stimulation

INTERVENTIONS:
Other: Comprehensive Intervention or Comprehensive Intervention Combined with Electrical vagus nerve stimulation — Comprehensive intervention includes multidisciplinary collaboration, screening and assessment, oral sensory training, oral motor training, respiratory training, and feeding management. Transcutaneous electrical stimulation of the vagus nerve at the lateral neck was performed by rehabilitation therapists. The cervical vagus nerve accompanies the carotid artery and is located at the groove between the trachea and the sternocleidomastoid muscle, which can be located by touching the carotid pulse. The two electrodes were pasted along the path of the cervical vagus nerve.
  Arms: Comprehensive Intervention Combined with Vagus Nerve Stimulation Group; Comprehensive Intervention Group

SUMMARY:
This study aims to establish a practical comprehensive intervention program for dysphagia after extubation in adult ICU patients based on the best evidence of its assessment and intervention, through expert panel discussion and Delphi method. In addition, combining the preliminary experimental results of vagus nerve stimulation applied to PED patients, we further develop a comprehensive intervention program for dysphagia after extubation based on neural regulation mechanism. Finally, the implementation effect of this PED comprehensive intervention program based on neural regulation mechanism will be verified through clinical application.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who met the diagnostic criteria of PED were changed to SSA score ≥24
2. aged from 18 to 90 years old;
3. oral or nasotracheal intubation for ≥48 hours;
4. Clear mind
5. Glasgow score ≥13 points, with good cooperation ability;
6. There was no contraindication to oral feeding after extubation

Exclusion Criteria:

1. Other diseases that affect swallowing function (such as stroke, Parkinson's disease, head and neck deformity, radiotherapy after head and neck cancer, burn with inhalation injury, esophageal cancer, chronic obstructive pulmonary disease, etc.);
2. history of reflux and aspiration;
3. tracheotomy;
4. isolation treatment due to respiratory infectious diseases;
5. the presence of implantable electronic devices (e.g., pacemakers, cochlear implants);
6. Traumatic vagus recurrent laryngeal nerve injury, history of vagus nerve surgery, or vagus nerve injury

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
functional oral intake scale（FOIS） | up to 90 days
  FOIS consists of seven levels: ① Score 1, unable to eat orally at all; ② Score 2, dependent on tube feeding, minimum attempt to eat food or liquid; ③ Score 3, dependent on tube feeding, taking single texture food or liquid orally; ④ Score 4, completely oral intake of single texture food; ⑤ score 5: fully oral intake of a variety of food textures, but with special preparation or compensation; ⑥6 points, completely oral feeding without special preparation, but with special food restriction; ⑦7 points, complete oral feeding without restriction, the higher the score, the better the swallowing function of the patient. In this study, a FOIS score of 6-7 was defined as full oral feeding
standardized Swallowing Assessment（SSA） | up to 90 days
  The first part is the clinical examination.The second part involves observing the patient's ability to swallow 5 mL of water, repeated three times. If there are no abnormalities detected in the above examinations, the amount of water for swallowing is then increased to 60 mL. To obtain the total score, the scores from all three parts are summed up.

SECONDARY OUTCOMES:
Rate of total oral feeding after the intervention | up to 90 days
  After the intervention, the patient's score on the Functional Oral Intake Scale (FOIS) was between 6 and 7, indicating that the patient has recovered the ability to eat orally.
Duration of Enteral Nutrition Tube Indwelling | up to 90 days
  The duration of the nasogastric tube or nasointestinal tube indwelling in the patient
Rate of Re-intubation after Endotracheal Intubation | up to 90 days
  The rate of re-intubation during the intervention period after extubation in patients who have undergone endotracheal intubation
Incidence of aspiration within one week after extubation | up to 90 days
  Incidence of aspiration within one week after extubation
The incidence of aspiration pneumonia within one week after extubation | up to 90 days
  The incidence of aspiration pneumonia within one week after extubation
Inflammation-related indicators: serum C-reactive protein (CRP) | up to 90 days
  Monitoring of patients' inflammatory marker
Inflammation-related indicators: serum interleukin-6 (IL-6) | up to 90 days
  Monitoring of patients' inflammatory marker
Inflammation-related indicators: serum procalcitonin, acetylcholine (ACh) | up to 90 days
  Monitoring of patients' inflammatory markers
Inflammation-related indicators: high mobility group box-1 protein (HMGB1) | up to 90 days
  Monitoring of patients' inflammatory marker
Days of ICU hospitalization | up to 90 days
  Days of ICU hospitalization
Total days of hospitalization | up to 90 days
  Total days of hospitalization
In-hospital survival rate | up to 90 days
  The number of patients who survive during hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Jinhua Municipal Central Hospital, Jinhua, China

IPD SHARING:
Plan to Share IPD: No